CLINICAL TRIAL: NCT06832683
Title: Comparison of the Efficacy of Intravenous Propofol-Ketamine and Sevoflurane Administered Via Face Mask in Children Undergoing Magnetic Resonance Imaging: A Prospective, Randomized, Parallel-Group Study
Brief Title: Efficacy of Propofol-Ketamine and Sevoflurane in Children Undergoing Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Bedirhan Günel, Medical Doctor, Kocaeli City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KSH-ANREA-BG-04
Record Dates: First submitted 2025-02-01; First posted 2025-02-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Recovery Period; Hypoxemia; Patient Safety
Keywords: recovery period; Hypoxemia; Patient Safety; Sedation, Moderate; propofol; ketamine; sevoflurane
MeSH Terms: conditions — Hypoxia; Lymphoma, Follicular | interventions — Sevoflurane; Propofol; Ketamine

STUDY DESIGN:
Intervention Model Description: A Prospective, Randomized, Parallel-Group Study
Who Masked: Participant
Masking Description: Only the participants will be blinded, making this a single-blind study design. The second anesthesiologist measuring the values in the PACU will also remain blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): Intravenous propofol and ketamine will be administered to the patients in this group.
  Interventions: Drug: Propofol; Drug: Ketamine
- Group S (Active Comparator): Sevoflurane will be administered via a procedural oxygen mask to the patients in this group.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — For Group S, 8% sevoflurane was administered for induction via the procedural oxygen mask for 2 minutes through the external output of the anesthesia machine. The concentration was then reduced to 2%. If any undesired movements occurred, they were recorded, and the sevoflurane concentration was increased by 0.5%.
  Other Names: Group S
  Arms: Group S
Drug: Propofol — In Group P, 1.0 mg/kg propofol as a bolus. In the event of undesired movements, an additional 0.5 mg/kg of propofol was administered, and all additional doses were recorded.
  Other Names: Group P
  Arms: Group P
Drug: Ketamine — In Group P, 1 mg/kg, single dose ketamine was administered intravenously and all additional doses were recorded.
  Other Names: Group P
  Arms: Group P

SUMMARY:
Magnetic resonance imaging (MRI) is becoming increasingly important in the diagnosis and follow-up of pediatric diseases. However, successful MRI requires complete and prolonged immobility, which can be challenging for young children and infants. To overcome this challenge, various anesthesia techniques are employed by anesthesiologists. The ideal anesthesia method for children during MRI should be both safe and enable rapid recovery, allowing the child to remain still during the procedure while minimizing risks during the recovery period.

**Sevoflurane has become a popular choice for this purpose due to its rapid onset, limited respiratory side effects at low concentrations, reduced airway irritation, and hemodynamic stability. However, propofol and ketamine, used as an alternative sedation method, are also being increasingly utilized during these procedures. The major side effects of propofol include respiratory depression, apnea, loss of protective reflexes, and hemodynamic instability. To minimize these side effects, some experts recommend the combined use of propofol and ketamine. This combination provides effective sedation while also contributing to a reduction in side effects.

In this context, the aim of our study is to compare the efficacy of intravenous propofol and ketamine with sevoflurane administered via a face mask during pediatric MRI.

DETAILED DESCRIPTION:
Participants were randomized in a 1:1 ratio using a computer program, stratified based on MRI durations, and divided into two groups: Group S and Group P.

All participants received intravenous midazolam at a dose of 0.05 mg/kg (max 2 mg). During MRI, all patients were monitored with pulse oximetry and end-tidal CO2, and procedural oxygen masks (POM) were applied to deliver oxygen at a flow rate of 5 L/min. For Group S, 8% sevoflurane was administered for induction via the procedural oxygen mask for 2 minutes through the external output of the anesthesia machine. The concentration was then reduced to 2%. If any undesired movements occurred, they were recorded, and the sevoflurane concentration was increased by 0.5%.

In Group P, 1 mg/kg ketamine was administered intravenously, followed by 1.0 mg/kg propofol as a bolus. In the event of undesired movements, an additional 0.5 mg/kg of propofol was administered, and all additional doses were recorded. The target sedation level was set at a Ramsay Sedation Scale (RSS) score of 4, which was maintained throughout the procedure. At the end of the procedure, patients were awakened with verbal and tactile stimulation. Once an RSS score of 2 was achieved, they were transferred to the Post-Anesthetic Care Unit (PACU).

Vital signs, procedure durations, and drug doses were recorded for each patient during the procedure. All clinical decisions regarding the patients were made by the attending anesthesiologist. In the PACU, patients with a modified Aldrete score of 10 were deemed eligible for discharge. After discharge approval, all patients were observed in the outpatient unit for 1 hour. The study concluded at this point.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3 months to 10 years.
* Classified as ASA I-II according to the American Society of Anesthesiologists (ASA) classification.
* Patients scheduled for MRI at Kocaeli City Hospital MRI unit.

Exclusion Criteria:

* Families or children who do not consent to participate in the study.
* Patients with allergies to ketamine, propofol, midazolam, or sevoflurane.
* Patients with known pulmonary or cardiac diseases.
* Patients with known congenital craniofacial or neck anomalies.
* Patients dependent on oxygen therapy.
* Patients with a recent respiratory tract infection within the past 2 weeks.
* Patients requiring tracheal intubation, laryngeal mask, or ventilator support.
* Patients at risk of upper airway obstruction.
* Patients with behavioral problems.
* Patients with gastroesophageal reflux disease.
* Patients with lethargy, stupor, or unresponsiveness to stimuli due to any cause
* Patients with active use of antiepileptic or antipsychotic medications

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Recovery time | From the end of the MRI scan until the patient reaches a Ramsay Sedation Scale (RSS) score of 2, assessed for a maximum of 60 minutes.
  Recovery time was defined as the duration (measured in minutes) from the end of the MRI scan until the patient reached a Ramsay Sedation Scale (RSS) score of 2. The Ramsay Sedation Scale ranges from 1 (awake) to 6 (deep sedation), with higher scores indicating deeper sedation. In this study, an RSS score of 2 was considered the criterion for sufficient recovery.

SECONDARY OUTCOMES:
Discharge time | From the completion of the procedure until the child's Modified Aldrete Score reaches 10, assessed for a maximum of 60 minutes.
  Discharge time was defined as the duration (measured in minutes) from the completion of the procedure until the child's Modified Aldrete Score reached 10, indicating readiness for discharge. The Modified Aldrete Score ranges from 0 to 10, with higher scores representing better recovery status. A score of 10 was considered the criterion for discharge readiness in this study.
Anesthesia duration | From the start of anesthesia induction to the completion of the MRI procedure, assessed for a maximum of 60 minutes.
  Anesthesia duration was defined as the time (measured in minutes) from the start of anesthesia induction until the completion of the MRI procedure.
Incidence of hypoxemia | Continuous SpO2 monitoring will be performed throughout the procedure]
  Incidence of hypoxemia during sedation (defined as SpO2 < 93%).
Number of hypoxemia episodes | Continuous SpO2 monitoring will be performed throughout the procedure
  a new episode was recorded if SpO2 fell below 93% again after reaching SpO2 ≥ 93% for at least 30 seconds
Duration of hypoxemia | Continuous SpO2 monitoring will be performed throughout the procedure
  defined as the time to reach SpO2 ≥ 93%
Minimum SpO2 | Continuous SpO2 monitoring will be performed throughout the procedure]
  observed during the procedure
airway management | Interventions related to airway management causing interruptions during the procedure
  Procedure interruptions due to airway interventions during the procedure (chin lift, jaw thrust, mask ventilation, need for suctioning).
Additional anesthetic intervention | during procedure
  Additional anesthetic intervention due to undesired movements disrupting image quality and causing interruptions in the procedure.
Image quality | immediately after the procedure
  Image quality was evaluated by a radiologist who was not involved in the imaging process, using a 10-point analog scale (0: unacceptable, 5: diagnosis not possible, 8: acceptable, 10: excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Bedirhan Günel, MD, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Bedirhan Günel, Kocaeli, İ̇zmi̇t, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal data and study data will not be shared.

REFERENCES:
- [Background] Schmitz A, Weiss M, Kellenberger C, O'Gorman Tuura R, Klaghofer R, Scheer I, Makki M, Sabandal C, Buehler PK. Sedation for magnetic resonance imaging using propofol with or without ketamine at induction in pediatrics-A prospective randomized double-blinded study. Paediatr Anaesth. 2018 Mar;28(3):264-274. doi: 10.1111/pan.13315. Epub 2018 Jan 27. PMID 29377404
- [Background] Ogurlu M, Orhan ME, Bilgin F, Sizlan A, Yanarates O, Yilmaz N. Efficacy of different concentrations of sevoflurane administered through a face mask for magnetic resonance imaging in children. Paediatr Anaesth. 2010 Dec;20(12):1098-104. doi: 10.1111/j.1460-9592.2010.03438.x. PMID 21199119